CLINICAL TRIAL: NCT07387796
Title: Clinical and Neurobehavioral Changes With GLP-1 (Glucagon-like Peptide-1) Discontinuation
Brief Title: Clinical and Neurobehavioral Changes With Weight Loss Drug Discontinuation and Reinitiation
Acronym: CLIN-GLP1
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Francesca Filbey, Professor, The University of Texas at Dallas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB-26-3
Record Dates: First submitted 2026-01-08; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Drug Discontinuation; Substance Use Disorders; Eating Behavior Changes; Tirzepatide
Keywords: Tirzepatide; Drug Discontinuation; Substance Use Disorders; Eating Behavior Changes
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Tirzepatide Discontinuation and Re-Initiation Arm (Experimental): Participants in this single-group arm will complete three study visits that occur while they are taking tirzepatide, during a 3-4 week pause from the medication, and after they restart tirzepatide for 6-8 weeks. All medication changes are supervised by a study physician. At each visit, participants will complete interviews, questionnaires, cognitive tasks, magnetic resonance imaging (MRI) brain scans, and provide stool samples. They will also complete two short check-in phone calls and an online BrainHealth Index assessment between visits.
  Interventions: Other: Discontinuation and Reinitiation of Tirzepatide

INTERVENTIONS:
Other: Discontinuation and Reinitiation of Tirzepatide — Participants will temporarily pause their tirzepatide medication for 3-4 weeks and then restart it for 6-8 weeks under the supervision of a study physician. The medication change is done only for research purposes to study how stopping and restarting tirzepatide affects brain activity, appetite, mood, and other health measures. During this period, participants will complete MRI scans, behavioral assessments, questionnaires, and provide stool samples across three study visits.

SUMMARY:
The goal of this clinical study with research procedures is to learn how stopping and restarting tirzepatide (a medication that helps regulate blood sugar and appetite) affects brain activity, behavior, and health in adults ages 18-70 who are currently taking tirzepatide. Specifically, the study aims to examine how a short pause in tirzepatide affects hunger, mood, sleep, and daily functioning; how stopping and restarting tirzepatide alters brain chemistry and brain responses to food-related images; and how these changes relate to health measures such as quality of life and emotional well-being. There is no comparison group; instead, researchers will assess changes within each participant across three time points: while taking tirzepatide, after stopping it for 3-4 weeks, and after restarting it for 6-8 weeks. Participants will attend three in-person visits lasting approximately 3-4 hours each, during which they will complete interviews, questionnaires, and cognitive tasks; provide a urine sample (pregnancy screening for females); undergo a brain scan using magnetic resonance imaging (MRI) and MR spectroscopy (MRS); and receive a kit to provide a small stool sample. Participants will also complete two brief check-in phone calls between visits and the online BrainHealth Index between sessions, which includes surveys and cognitive tasks. All changes to tirzepatide use will occur under the supervision of a study physician to support participant safety and comfort, and the total study duration is approximately 13 weeks.

DETAILED DESCRIPTION:
This study specifically recruits individuals currently being prescribed for tirzepatide. The experimental design will consist of a brief discontinuation of the drug for roughly 3-4 weeks followed by a reinitiation of the medication. Prescription and administration of tirzepatide is done as part of normal patient care and is not a component of the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years.
* Currently on tirzepatide.
* Currently receiving care from University of Texas- Southwestern (UTSW) Weight Wellness Clinic.
* Cognitively capable of understanding and signing informed consent.
* Be proficient in English.

Exclusion Criteria:

* History of major neurological or psychiatric disorders, including substance use disorders that might confound brain imaging results (e.g., stroke, epilepsy, multiple sclerosis, schizophrenia, major depression requiring hospitalization).
* Diagnosis of Type 2 Diabetes.
* Use of medications affecting weight other than tirzepatide.
* Pregnancy or breastfeeding.
* MR contraindications:
* Heart pacemaker, heart valve replacement, or aortic clips
* Metal fragments in the eyes, skin, or elsewhere in the body
* Brain clips or pieces of metal used in aneurysm surgery or intercranial bypass
* Venous umbrella
* Pieces of metal in the body resulting from work as a sheet-metal worker or welder
* Clips placed in an internal organ
* Prosthetic devices, such as middle ear, eye, joint, or penile implants
* Joint replacement
* Hearing aid that cannot be removed
* Neurostimulator
* Insulin pump
* Shunts or stents
* Metal mesh or coil implants
* Metal plate, pin, screws, or wires, or any other metal implants

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change From On-Treatment to Discontinuation and Re-Initiation in Food Cue-Evoked BOLD Response in Reward and Salience Brain Regions | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measures within-participant change in blood-oxygen-level-dependent (BOLD) signal during a food cue reactivity task, assessed using functional magnetic resonance imaging (fMRI).
  BOLD response will be quantified as the mean percent signal change in predefined reward- and salience-related regions of interest (including the ventral striatum and insula) during food image presentation relative to non-food control images. Higher BOLD values indicate greater neural responsivity to food cues.

SECONDARY OUTCOMES:
Change From Baseline in Resting-State Functional Connectivity Within Salience and Executive Control Networks | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measures within-participant change in resting-state functional connectivity, assessed using fMRI. Connectivity strength will be calculated using correlation coefficients between predefined brain regions within salience and executive control networks. Higher values indicate stronger functional connectivity.
Change From Baseline in Brain Neuromelanin Signal | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in neuromelanin signal intensity in the substantia nigra. Neuromelanin-sensitive magnetic resonance imaging (MRI) will be used to quantify signal intensity within a predefined substantia nigra region of interest. Higher values indicate greater neuromelanin-related signal intensity.
Change From Baseline in Brain Glutamate Levels | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measures within-participant change in neurochemical and dopaminergic markers associated with reward processing. Glutamate levels will be measured in the medial prefrontal cortex using magnetic resonance spectroscopy (MRS). Higher values indicate greater metabolite concentration or signal intensity.
Change From Baseline in State Food Craving Severity | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in momentary food craving severity. Food cravings will be measured using the Food Cravings Questionnaire-State (FCQ-S), a self-report instrument assessing current craving intensity. Scores range from 15 to 75, with higher scores indicating greater food craving severity.
Change From Baseline in Trait Food Craving Severity. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in habitual food craving frequency and intensity. Trait-level food cravings will be assessed using the Food Cravings Questionnaire-Trait, a self-report questionnaire. Scores range from 39 to 234, with higher scores indicating more frequent and intense food cravings.
Change From Baseline in Addictive-Like Eating Symptoms. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in addictive-like eating behaviors. Addictive-like eating symptoms will be assessed using the Yale Food Addiction Scale 2.0, a self-report measure of addictive-like eating based on diagnostic criteria. Symptom counts range from 0 to 11, with higher scores indicating greater severity of addictive-like eating behavior.
Change From Baseline in Intrusive Food-Related Thoughts. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in the frequency of intrusive food-related thoughts. Intrusive food-related cognitions will be assessed using the Food Noise Questionnaire, a self-report measure consisting of five items assessing persistent and intrusive thoughts about food. Total scores range from 0 to 20, with higher scores indicating greater food noise and more frequent intrusive food-related thoughts.
Change From Baseline in Dietary Pattern Quality. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in dietary behaviors and overall eating patterns. Dietary patterns will be assessed using the Rapid Eating Assessment for Participants - Shortened Version, a self-report questionnaire evaluating habitual dietary behaviors. Total scores range from 13 to 39, with higher scores indicating poorer dietary patterns.
Change From Baseline in Attentional Bias Toward Food Cues. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in attentional bias toward food-related stimuli. Attentional bias will be assessed using a Food-Modified Stroop Task, a performance-based behavioral task. Attentional bias is quantified as the difference in reaction time (milliseconds) between food-related and neutral stimuli. Greater reaction time differences indicate stronger attentional bias toward food cues.
Change From Baseline in Perceived Loss of Control Over Eating. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in perceived loss of control over eating behavior. Perceived loss of control will be assessed using the Loss of Control Over Eating Scale-Short Form, a self-report questionnaire assessing the subjective experience of being unable to control eating. Total scores range from 0 to 28, with higher scores indicating greater perceived loss of control over eating.
Change From Baseline in Psychological Responsiveness to Food Availability. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in psychological responsiveness to the food environment. Responsiveness to food availability will be assessed using the Power of Food Scale, a self-report questionnaire measuring the psychological impact of food availability independent of actual consumption. Scores are calculated as a mean item score ranging from 1 to 5, with higher scores indicating greater psychological impact of food availability.
Change From Baseline in Uncontrolled Eating Behavior. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in uncontrolled eating behavior. Uncontrolled eating will be assessed using the Uncontrolled Eating subscale of the Three-Factor Eating Questionnaire, a self-report measure of tendencies toward loss of control over eating. Subscale scores range from 0 to 36, with higher scores indicating poorer regulation of eating behavior.
Change From Baseline in Mood Disturbance. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in mood disturbance. Mood will be assessed using the Profile of Mood States-Second Edition, a validated self-report questionnaire assessing multiple mood domains including tension, depression, anger, vigor, fatigue, and confusion. Mood disturbance will be quantified using the Total Mood Disturbance score, which ranges from -32 to 200, with higher scores indicating greater overall mood disturbance (reflecting higher negative mood and lower vigor).
Change From Baseline in Perceived Stress. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in perceived psychological stress. Perceived stress will be measured using the Perceived Stress Scale (PSS), a self-report questionnaire assessing the degree to which situations in one's life are appraised as stressful over the past month. Scores range from 0 to 40, with higher scores indicating greater perceived stress.
Change From Baseline in Emotional Health and Psychological Well-Being. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in emotional health and psychological well-being. Emotional functioning will be assessed using the NIH Toolbox Emotion Battery, a self-report assessment comprising multiple domains, including negative affect, psychological well-being, stress and self-efficacy, and social relationships. Domain scores are reported as standardized T-scores (mean = 50, standard deviation = 10; typical range ~20-80). For negative affect domains, higher scores indicate worse emotional health, whereas for well-being and social functioning domains, higher scores indicate better emotional health.
Change From Baseline in Quality of Life. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in quality of life. Quality of life will be assessed using the World Health Organization Quality of Life-BREF, a 26-item self-report questionnaire assessing perceived quality of life across physical health, psychological health, social relationships, and environmental domains. Total scores range from 26 to 130, with higher scores indicating better overall quality of life.
Change From Baseline in Withdrawal-Related Psychological Symptoms. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in withdrawal-related psychological and behavioral distress during tirzepatide discontinuation. Withdrawal symptoms will be assessed using a Withdrawal Symptom Checklist, a self-report questionnaire assessing appetite and physiological symptoms, eating behavior and perceived control, restrictive dieting and compensatory behaviors, mood and emotional distress, and general physical and functional impairment associated with medication withdrawal. Items are rated on a 5-point scale ranging from 0 (not at all/never) to 4 (very severe/very often) and summed to create a total score. Total scores range from 0 to 128, with higher scores indicating greater withdrawal-related psychological and behavioral distress.
Change From Baseline in Sleep Quality as Measured by the Pittsburgh Sleep Quality Index | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  The Pittsburgh Sleep Quality Index (PSQI) is a 19-item self-report questionnaire assessing subjective sleep quality over the past month. Global scores range from 0 to 21, with higher scores indicating poorer sleep quality.
Change From Baseline in Addiction-Related Problem Severity | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in addiction-related problem severity across multiple functional domains. Addiction-related severity will be assessed using the Addiction Severity Index, a standardized semi-structured interview administered by trained study personnel. The Addiction Severity Index evaluates seven domains: medical status, employment/support status, alcohol use, drug use, legal status, family/social functioning, and psychological status, based on both past 30-day functioning and lifetime history. Domain-specific composite scores range from 0 to 1, with higher scores indicating greater addiction-related problem severity.
Change From Baseline in Substance Use Frequency and Quantity. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in substance use behavior. Substance use frequency and quantity will be measured using the Timeline Follow-Back (TLFB) method, which captures the number of days and amount of alcohol, nicotine, and cannabis use over the past 30 days. Higher values indicate more frequent or greater substance use.
Change From Baseline in Risky and Impulsive Behavior. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in engagement in risky, impulsive, and self-destructive behaviors. Behaviors will be assessed using the Risky, Impulsive, and Self-Destructive Behavior Questionnaire, a 38-item self-report measure. Frequency responses are binned and summed to create a total score ranging from 0 to 152, with higher scores indicating greater engagement in risky, impulsive, and self-destructive behaviors.

OTHER OUTCOMES:
Change From Baseline in Gut-Derived Neurotransmitter Levels. | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in gut-derived neurotransmitter levels associated with tirzepatide discontinuation and re-initiation. Neurotransmitter levels will be measured from stool samples collected at each study timepoint and analyzed for gut-derived neurotransmitters relevant to brain-gut signaling. Changes in values reflect alterations in gut-derived neurotransmitter levels.
Change From Baseline in Gut Microbiome and Inflammatory Marker Profiles | Baseline (on tirzepatide), 3-4 weeks of discontinuation, and 6-8 weeks of re-initiation
  This outcome measure assesses within-participant change in gut microbiome composition and gut-related inflammatory markers. Exploratory analyses will be conducted on stool samples to evaluate changes in microbial profiles and inflammatory markers associated with tirzepatide discontinuation and re-initiation. Higher or lower values reflect changes depending on the specific marker assessed.
Change in Multidimensional Brain Health as Measured by the BrainHealth Index | Between baseline and discontinuation (about 2 weeks after baseline), and between discontinuation and re-initiation (about 4 weeks after start of reinitiation)
  This outcome measure assesses within-participant change in overall brain health using the BrainHealth Index (BHI), a multidimensional composite derived from standardized self-report questionnaires and objective cognitive performance measures developed at the Center for BrainHealth. The BHI integrates measures across three domains: cognitive function/clarity (e.g., attention, learning and memory, reasoning, processing speed, and sleep quality), emotional balance (e.g., mood, stress, anxiety, happiness), and social connectedness (e.g., compassion, social support, resilience, engagement in meaningful activities, and life satisfaction). Component measures are standardized and combined using predefined BrainHealth Index aggregation procedures to generate a single composite score, with higher scores indicating better overall brain health.
Occurrence and Severity of Withdrawal-Related Symptoms During Medication Discontinuation | Between baseline and discontinuation (about 2 weeks after baseline), and between discontinuation and re-initiation (about 4 weeks after start of re-initiation)
  This outcome measure assesses within-participant change in withdrawal-related symptom severity during tirzepatide discontinuation. Withdrawal symptoms will be assessed using the Glucagon-like Peptide-1 (GLP-1) Withdrawal Symptom Checklist Brief Version, a self-report questionnaire assessing appetite and physiological symptoms, eating behavior and loss of control, restrictive dieting and compensatory behaviors, psychological/mood distress, and general physical and functional symptoms over the past 7 days. Items are rated on a 5-point scale ranging from 0 (not at all/never) to 4 (very severe/very often). A total symptom severity score is calculated as the mean of items 1-5, yielding a minimum score of 0 and a maximum of 4, with higher scores indicating greater withdrawal-related symptom severity. An additional item assessing overall subjective burden is collected separately for descriptive purposes on a scale of 0 to 4 with higher scores indicating higher burden.

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Filbey, Doctor of Philosophy, Principal Investigator — The University of Texas at Dallas
Locations (1):
- Center for BrainHealth, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jurca R, Jackson AS, LaMonte MJ, Morrow JR, Blair SN, Wareham NJ, et al. Assessing cardiorespiratory fitness without performing exercise testing. Am J Prev Med. (2005) 29:185-93. doi: 10.1016/j.amepre.2005.06.00
- [Background] Burckhardt CS, Anderson KL. The quality of life scale (QOLS): reliability, validity, and utilization. Health Qual Life Outcomes. (2003) 1:60. doi: 10.1186/1477-7525-1-60
- [Background] Connor KM, Davidson JRT. Development of a new resilience scale: the Connor-Davidson Resilience Scale (CD-RISC). Depress Anxiety. (2003) 18:76-82. doi: 10.1002/da.10113
- [Background] Sherbourne CD, Stewart AL. The MOS social support survey. Soc Sci Med. (1991) 32:705-14. doi: 10.1016/0277-9536(91)90150-b
- [Background] Hills P, Argyle M. The Oxford Happiness Questionnaire: a compact scale for the measurement of psychological well-being. Pers Indiv Differ. (2002) 33:1073-82. doi: 10.1016/S0191-8869(01)00213-6
- [Background] Eakman AM. Convergent validity of the engagement in meaningful activities survey in a college sample. OTJR. (2011) 30:23-32. doi: 10.3928/15394492-20100122-02
- [Background] Lovibond PF, Lovibond SH. The structure of negative emotional states: comparison of the Depression Anxiety Stress Scales (DASS) with the beck depression and anxiety inventories. Behav Res Ther. (1995) 33:335-43. doi: 10.1016/0005-7967(94)00075-u
- [Background] Strauss C, Lever Taylor B, Gu J, Kuyken W, Baer R, Jones F, et al. What is compassion and how can we measure it? A review of definitions and measures. Clin Psychol Rev. (2016) 47:15-27. doi: 10.1016/j.cpr.2016.05.004
- [Background] Johnson LKD. The Light Triad Scale: developing and validating a preliminary measure of prosocial orientation (Master's thesis). [Electronic Thesis and Dissertation Repository: 5515], The University of Western Ontario (2018). Available online at: https://ir.lib.uwo.ca/etd/551
- [Background] Vas AK, Chapman SB, Cook LG (editors). Language impairments in traumatic brain injury: a window into complex cognitive performance. In: Handbook of Clinical Neurology: Traumatic Brain Injury Part II. Amsterdam: Elsevier (2015). p. 497-510
- [Background] Hanten G, Li X, Chapman SB, Swank P, Gamino J, Roberson G, et al. Development of verbal selective learning. Dev Neuropsychol. (2007) 32:585-96. doi: 10.1080/87565640701361112
- [Background] Zhang, X., Wang, H., Kilpatrick, L. A., Dong, T. S., Gee, G. C., Labus, J. S., Osadchiy, V., Beltran-Sanchez, H., Wang, M. C., Vaughan, A., & Gupta, A. (2023). Discrimination exposure impacts unhealthy processing of food cues: Crosstalk between the brain and gut. Nature Mental Health, 1(11), 841-852. https://doi.org/10.1038/s44220-023-00134-9
- [Background] Vartanian, M., Jahanitabesh, A., Christensen, J. F., Staub, H., Jensen, D. E. A., Villringer, A., & Witte, A. V. (2025). Neural responses to visual food cues according to weight and hunger state: A systematic review and meta-analysis. Neuroscience and Biobehavioral Reviews, 177, 106301. https://doi.org/10.1016/j.neubiorev.2025.106301
- [Background] The WHOQOL Group. (1994). The Development of the World Health Organization Quality of Life Assessment Instrument (the WHOQOL). In J. Orley & W. Kuyken (Eds.), Quality of Life Assessment: International Perspectives (pp. 41-57). Springer Berlin Heidelberg. https://doi.org/10.1007/978-3-642-79123-9_4
- [Background] Stunkard, A. J., & Messick, S. (1985). The three-factor eating questionnaire to measure dietary restraint, disinhibition and hunger. Journal of Psychosomatic Research, 29(1), 71-83. https://doi.org/10.1016/0022-3999(85)90010-8
- [Background] Sobell, L. C., & Sobell, M. B. (1992). Timeline Follow-Back. In R. Z. Litten & J. P. Allen (Eds.), Measuring Alcohol Consumption (pp. 41-72). Humana Press. https://doi.org/10.1007/978-1-4612-0357-5_3
- [Background] Segal-Isaacson, C. J., Wylie-Rosett, J., & Gans, K. M. (2004). Validation of a Short Dietary Assessment Questionnaire: The Rapid Eating and Activity Assessment for Participants Short Version (REAP-S). The Diabetes Educator, 30(5), 774-781. https://doi.org/10.1177/014572170403000512
- [Background] Sadeh, N., & Baskin-Sommers, A. (2017). Risky, Impulsive, and Self-Destructive Behavior Questionnaire (RISQ): A Validation Study. Assessment, 24(8), 1080-1094. https://doi.org/10.1177/1073191116640356
- [Background] Rejeski, W. J., Burdette, J., Burns, M., Morgan, A. R., Hayasaka, S., Norris, J., Williamson, D. A., & Laurienti, P. J. (2012). Power of food moderates food craving, perceived control, and brain networks following a short-term post-absorptive state in older adults. Appetite, 58(3), 806-813. https://doi.org/10.1016/j.appet.2012.01.025
- [Background] Nijs, I. M. T., Franken, I. H. A., & Muris, P. (2007). The modified Trait and State Food-Cravings Questionnaires: Development and validation of a general index of food craving. Appetite, 49(1), 38-46. https://doi.org/10.1016/j.appet.2006.11.001
- [Background] McLELLAN, A. T., Luborsky, L., Woody, G. E., & O??Brien, C. P. (1980). An Improved Diagnostic Evaluation Instrument for Substance Abuse Patients: The Addiction Severity Index. The Journal of Nervous and Mental Disease, 168(1), 26-33. https://doi.org/10.1097/00005053-198001000-00006
- [Background] Latner, J. D., Mond, J. M., Kelly, M. C., Haynes, S. N., & Hay, P. J. (2015). Loss of Control Over Eating Scale. In T. Wade (Ed.), Encyclopedia of Feeding and Eating Disorders (pp. 1-4). Springer Singapore. https://doi.org/10.1007/978-981-287-087-2_5-1
- [Background] Heuchert, J. P., & McNair, D. M. (2012). Profile of Mood States 2nd EditionTM [Dataset]. https://doi.org/10.1037/t05057-000
- [Background] Gearhardt, A. N., Corbin, W. R., & Brownell, K. D. (2016). Development of the Yale Food Addiction Scale Version 2.0. Psychology of Addictive Behaviors: Journal of the Society of Psychologists in Addictive Behaviors, 30(1), 113-121. https://doi.org/10.1037/adb0000136
- [Background] Flint, A., Raben, A., Blundell, J., & Astrup, A. (2000). Reproducibility, power and validity of visual analogue scales in assessment of appetite sensations in single test meal studies. International Journal of Obesity, 24(1), 38-48. https://doi.org/10.1038/sj.ijo.0801083
- [Background] Diktas, H. E., Cardel, M. I., Foster, G. D., LeBlanc, M. M., Dickinson, S. L., Ables, E. M., Chen, X., Nathan, R., Shapiro, D., & Martin, C. K. (2025). Development and validation of the Food Noise Questionnaire. Obesity (Silver Spring, Md.), 33(2), 289-297.
- [Background] Davidson, E. J., & Wright, P. (2002). Selective processing of weight- and shape-related words in bulimia nervosa. Eating Behaviors, 3(3), 261-273. https://doi.org/10.1016/S1471-0153(02)00064-8
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Chapman, S. B., Fratantoni, J. M., Robertson, I. H., D'Esposito, M., Ling, G. S. F., Zientz, J., Vernon, S., Venza, E., Cook, L. G., Tate, A., & Spence, J. S. (2021). A Novel BrainHealth Index Prototype Improved by Telehealth-Delivered Training During COVID-19. Frontiers in Public Health, 9, 641754. https://doi.org/10.3389/fpubh.2021.641754
- [Background] Buysse, D. J., Reynolds, C. F., Monk, T. H., Berman, S. R., & Kupfer, D. J. (1989). The Pittsburgh sleep quality index: A new instrument for psychiatric practice and research. Psychiatry Research, 28(2), 193-213. https://doi.org/10.1016/0165-1781(89)90047-4
- [Background] Blechert, J., Meule, A., Busch, N. A., & Ohla, K. (2014). Food-pics: An image database for experimental research on eating and appetite. Frontiers in Psychology, 5. https://doi.org/10.3389/fpsyg.2014.00617
- [Background] Babakhanyan, I., McKenna, B. S., Casaletto, K. B., Nowinski, C. J., & Heaton, R. K. (2018). National Institutes of Health Toolbox Emotion Battery for English- and Spanish-speaking adults: Normative data and factor-based summary scores. Patient Related Outcome Measures, Volume 9, 115-127. https://doi.org/10.2147/PROM.S151658